CLINICAL TRIAL: NCT00962117
Title: Food Reinforcement Genotype Interactions and Eating
Brief Title: Relationship Between Dopamine Genetics, Food Reinforcement, Energy Intake and Obesity
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, SUNY Distinguished Professor of Pediatrics and Social and Preventive Medicine, State University of New York at Buffalo
Other Study IDs: 1066937; 1066937-1-44786
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Food Reinforcement; Energy Intake; Obesity; Dopamine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva DNA samples will be collected from all participants
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese/Non-obese

SUMMARY:
The purpose of the study is to determine whether the presentation of various foods produces an increase or decrease in responses on a motivational computer task. In addition, the study determines if energy intake or motivation to obtain food is related to the dopamine receptor genotype.

DETAILED DESCRIPTION:
One of the most important research areas in obesity is developing a better understanding of individual differences in factors that influence excess energy intake and positive energy balance. One key to understanding these individual differences is determining what factors underlie the motivation to eat. We have demonstrated in a series of studies that obese adults and children are more motivated to work for palatable, favorite foods than leaner peers and that those high in food reinforcement consume more food in an ad libitum eating task than those who do not find food as reinforcing. Dopamine (DA) is one of the major neurotransmitters involved in establishing the reinforcing value of food, and low levels of dopamine activity and a reduction in the number of DA receptors is associated with obesity. The general aim of the proposed research is to build upon this research to examine relationships between food reinforcement, obesity, and polymorphisms of genes within the dopaminergic system.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* 18-50 years of age
* No known eating disorder
* Moderate liking for study foods
* No current diagnosis of psychiatric disorder (e.g., anxiety or depression)
* Not on medications that would interfere with appetite (e.g., methylphenidate) or dopaminergic activity
* Non-diabetics

Exclusion Criteria:

* Smoker
* Pregnant women
* Current diagnosis of a psychiatric or eating disorder
* Dietary restrictions that would interfere with participation
* On medications that could interfere with appetite or olfactory responsiveness or use of antidepressants or any medication or dietary supplement that could affect appetite or dopaminergic activity
* Excessive use of alcohol (>21 drinks/week), alcoholism,current addiction to opiates, cocaine or stimulants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from newspaper ads, posters on campus and in community settings, web based recruitment (ads on Craig's list and on the department's website) and direct mail targeted to community residents between 18-50 years of age.
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard H Epstein, Ph.D., Principal Investigator — SUNY Buffalo

REFERENCES:
- [Derived] Lin H, Carr KA, Fletcher KD, Epstein LH. Food reinforcement partially mediates the effect of socioeconomic status on body mass index. Obesity (Silver Spring). 2013 Jul;21(7):1307-12. doi: 10.1002/oby.20158. Epub 2013 Jun 11. PMID 23754824
- [Derived] Epstein LH, Carr KA, Lin H, Fletcher KD, Roemmich JN. Usual energy intake mediates the relationship between food reinforcement and BMI. Obesity (Silver Spring). 2012 Sep;20(9):1815-9. doi: 10.1038/oby.2012.2. Epub 2012 Jan 13. PMID 22245983
- [Derived] Epstein LH, Lin H, Carr KA, Fletcher KD. Food reinforcement and obesity. Psychological moderators. Appetite. 2012 Feb;58(1):157-62. doi: 10.1016/j.appet.2011.09.025. Epub 2011 Oct 8. PMID 22005184
- [Derived] Epstein LH, Carr KA, Lin H, Fletcher KD. Food reinforcement, energy intake, and macronutrient choice. Am J Clin Nutr. 2011 Jul;94(1):12-8. doi: 10.3945/ajcn.110.010314. Epub 2011 May 4. PMID 21543545